CLINICAL TRIAL: NCT04991636
Title: Analysis of Respiration-induced Deformations in Visceral and Renal Arteries Before and After Stenting During Branched Stent Treatment.
Acronym: BEVAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A00911-40
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Complex Aortic Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protocol (Experimental): Each patient agreeing to participate in the study will be distributed in the protocol group and will receive an angioscan according to the protocol in pre-operative and at the usual post-operative check-up within 3 months after the operation. The usual procedure, foresees an angioscanner with injection of contrast product and the measurement of the images is performed during a deep breath. In order to obtain a complete respiratory cycle, the study procedure foresees in addition to the usual procedure, an image measurement during a deep exhalation.
  Interventions: Procedure: Angioscan

INTERVENTIONS:
Procedure: Angioscan — La procédure d'étude prévoit de prendre des images pendant une inspiration profonde ainsi que pendant une expiration profonde. Cette deuxième mesure ne nécessite pas l'administration d'une quantité supplémentaire de produit de contraste. Cependant, le temps d'exposition aux rayonnements ionisants est doublé. L'examen utilise une acquisition hélicoïdale en mode rapide. La durée de l'hélice est de l'ordre de 2 secondes en phase d'inspiration, puis il y a un délai de 5 secondes de machine (" demi-tour ") et à nouveau 2 secondes d'exposition en phase d'expiration, soit 4 secondes d'exposition effective aux rayonnements ionisants, le temps de la prise d'image et 9 secondes le temps total de l'examen. l'image et 9 secondes la durée totale de l'examen.

SUMMARY:
Aneurysm of the abdominal aorta is defined by a loss of parallelism of the arterial wall. The main risk of this pathology is the rupture of the aneurysm which is life threatening and this risk increases with the size of the aneurysm. Connected stents allow the management of complex thoracoabdominal aneurysms in patients at high surgical risk and/or contraindicated for open surgery. These endovascular techniques have demonstrated their safety and efficacy, however, long-term CT follow-up remains essential to detect complications such as endo-leaks and restenosis/thrombosis of visceral and renal stents. The prognostic factors of these complications remain poorly elucidated. The type of stent to be used could be an explanation, however, no stent has been proven to be superior in this application to date. Data from the literature suggest an influence of stents on the aortic geometry and the arterial axes of the digestive tract during respiratory movements. The work of the Stanford vascular surgery team shows that the deformations and modifications of the geometry of these stents induced by the respiratory cycle could have a negative impact by migration, stenosis and thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* no contre indication for coroscanner

Exclusion Criteria:

* pregnant woman
* allergy to iodinated contrast media
* vulnerable people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-09-07 (Estimated)

PRIMARY OUTCOMES:
Geometry of the visceral and renal branches | 1 day
  An angioscanner will be performed with injection in inspiration and expiration (breathing cycle) before and after stent placement for a fenestrated aortic endografts After reconstruction of a 3D volume of the aorta and extraction of the central lines of the different target arteries, the angle of the different visceral and renal branches will be measured during the respiratory cycle (inspiration; expiration) and compared before and after stenting.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France